CLINICAL TRIAL: NCT05375630
Title: Effects Vitamin K2 on Muscle Mass and Function in People With Muscle Weakness and Type 2 Diabetes
Brief Title: Vitamin K2 and Muscle Weakness in Type 2 Diabetes
Acronym: SARK2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dasman Diabetes Institute (Other)
Collaborators: Kappa Bioscience (Unknown)
Responsible Party: Principal Investigator, Dr. Ebaa Al Ozairi, Chief Medical Officer, Dasman Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA HM-2021-015
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Diabete Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vitamin K 2

STUDY DESIGN:
Intervention Model Description: Parallel Group Randomised Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): micro-crystalline cellulose placebo (one 380 mg tablet per day)
  Interventions: Dietary Supplement: Placebo
- Vitamin K2 (Active Comparator): micro-crystalline cellulose (one 380 mg tablet per day) where vitamin K2 (K2VITAL® 0.2% DELTA powder) is mixed into the formulation to a final vitamin K2 concentration of 240 μg/tablet
  Interventions: Dietary Supplement: Vitamin K2

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo
  Arms: Placebo
Dietary Supplement: Vitamin K2 — Vitamin K2
  Arms: Vitamin K2

SUMMARY:
The aim of the current study is to determine the effects of vitamin K2 supplementation on muscle size and function in adults with muscle weakness and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Physician confirmed type 2 diabetes.
* Age >/= 40 years
* No changes in anti-diabetic medication in the last 3 months.
* Muscle weakness (grip strength <27kg and females <16kg)

Exclusion Criteria:

* BMI of 45 or higher
* BP of 160/100mmHg or higher
* Cancer or cancer that has been in remission <5 years
* Any medical condition that prevents participants from exercising safely
* On anticoagulant therapy
* Currently consuming vitamin K2 supplements
* Current smoker

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Grip Strength | Baseline to one year
  Change in Grip Strength

SECONDARY OUTCOMES:
SPPB | Baseline to one year
  Change in Short Performance Physical Battery Test
HbA1c | Baseline to one year
  Change in glycated haemoglobin
Blood Pressure | Baseline to one year
  Change in blood pressure
Body Mass | Baseline to one year
  Change in body mass
Lean Mass | Baseline to one year
  Change in lean mass
Body Fat | Baseline to one year
  Change in body fat
BMC | Baseline to one year
  Change in bone mineral content
BMD | Baseline to one year
  Change in bone mineral density
Vitamin K status | Baseline to one year
  Change in vitamin K status

CONTACTS AND LOCATIONS:
Overall Officials: Ebaa AlOzairi, Principal Investigator — Dasman Diabetes Institute
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait